CLINICAL TRIAL: NCT06081699
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of a Single Oral Dose of TNP-2198 Capsules in Healthy Participants and the Effect of Food on the Pharmacokinetics of TNP-2198 Capsules in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effect of TNP-2198 Capsules After Single Oral Dose in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2198-01
Record Dates: First submitted 2023-09-22; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Single Ascending Doses Cohort 1 (Experimental): TNP-2198 Capsules 50mg
  Interventions: Drug: TNP-2198
- Single Ascending Doses Cohort 2 (Experimental): TNP-2198 Capsules 100mg
  Interventions: Drug: TNP-2198
- Single Ascending Doses Cohort 3 (Experimental): TNP-2198 Capsules 200mg
  Interventions: Drug: TNP-2198
- Single Ascending Doses Cohort 4 (Experimental): TNP-2198 Capsules 400mg
  Interventions: Drug: TNP-2198
- Single Ascending Doses Cohort 5 (Experimental): TNP-2198 Capsules 600mg
  Interventions: Drug: TNP-2198
- Single Ascending Doses Cohort 6 (Experimental): TNP-2198 Capsules 800mg
  Interventions: Drug: TNP-2198
- Single Ascending Doses Cohort 7 (Experimental): TNP-2198 Capsules 1000mg
  Interventions: Drug: TNP-2198
- Food Effect Cohort 8 (Experimental): TNP-2198 Capsules 200mg
  Interventions: Drug: TNP-2198
- Placebo Cohort 9 (Placebo Comparator): Placebo
  Interventions: Drug: TNP-2198 Placebo

INTERVENTIONS:
Drug: TNP-2198 — Oral
  Other Names: Rifasutenizol
  Arms: Food Effect Cohort 8; Single Ascending Doses Cohort 1; Single Ascending Doses Cohort 2; Single Ascending Doses Cohort 3; Single Ascending Doses Cohort 4; Single Ascending Doses Cohort 5; Single Ascending Doses Cohort 6; Single Ascending Doses Cohort 7
Drug: TNP-2198 Placebo — The placebo for TNP-2198 active drug
  Arms: Placebo Cohort 9

SUMMARY:
This was a single-center, randomized, double-blind, placebo-controlled phase 1 study to evaluate the safety, tolerability, pharmacokinetics of single ascending dose and the food effect on the pharmacokinetics of TNP-2198 capsules after single dose oral administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Those signed the informed consent form and fully understood the study contents, process and possible adverse reactions before participation in the study;
* Those are able to complete the study according to the requirements of the study protocol;
* Those (including the partner) are willing to use effective contraceptives from the screening up to 6 months after the last dose of study drug;
* Male and female subjects aged 18 to 55 years (inclusive);
* Male subjects no less than 50 kg and female subjects no less than 45 kg. BMI (Body Mass Index= body weight (kg)/height^2 (m^2)): 18-28kg/m^2 (inclusive);
* Health status: no clinically significant history of heart, liver, kidney, digestive tract, nervous system, respiratory system diseases, mental disorders or metabolic abnormalities;
* Normal results or abnormal results without clinical significance in physical examinations and vital signs;
* Clinical laboratory test results are within normal limits or abnormal but without clinical significance as judged by the investigator.

Exclusion Criteria:

* Average daily consumption of more than 5 cigarettes within 3 months before the study;
* History of hypersensitivity to study drug or its excipients, or allergic constitution (allergy to multiple drugs and food);
* History of drug and/or alcohol abuse (mean consumption of ≥ 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine);
* Blood donation or massive blood loss (> 450 mL) within 3 months prior to screening;
* Using any drug that changes liver enzyme activity within 28 days prior to screening;
* Using any prescription drug, over-the-counter drug, any vitamin product, or herbal medicine within 14 days prior to screening;
* Taking special diet (including dragon fruit, mango, grapefruit, etc.) or strenuous exercise, or having other factors that affect drug absorption, distribution, metabolism, excretion, etc., within 2 weeks prior to screening;
* Significant changes in diet or exercise habits recently;
* Taking other study drugs or participating in other clinical studies within 3 months before taking the study drug;
* With difficulty in swallowing or history of any gastrointestinal diseases that affect drug absorption;
* With any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers;
* Unable to tolerate standardized meal (two boiled eggs, one butter bacon toast, one box of fried potato chips, and one cup of whole milk) (only for subjects participating in the food effect study);
* With clinically significant ECG abnormalities;
* Female subjects who are lactating or have positive serum pregnancy result during the screening period, or have positive serum pregnancy result during the study;
* With symptoms or previous history of cardiovascular, digestive, respiratory, urinary, neurological, hematologic, immunological, endocrine system diseases, tumor, or psychiatric diseases;
* Clinically significant abnormalities in clinical laboratory tests, or other clinically significant findings (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, psychiatric, or cardiovascular disease);
* Positive viral hepatitis (including hepatitis B and C), HIV antibody, treponema pallidum antibody;
* Acute illness or concomitant medication from the time of signing informed consent to the time of study medication;
* Intake of chocolate, any caffeine- or xanthine-containing food or drink within 48 hours prior to administration of study drug;
* Intake of any alcohol-containing products within 48 hours prior to administration of study drug;
* Positive urine drug screening or history of drug abuse or drug addiction within the past 5 years;
* Other conditions that, in the opinion of the investigator, make the patient participating in this study inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Day 1 to Day 4
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) | Hour 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 after administration.
  Plasma concentrations of TNP-2198 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2198 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area Under the Plasma Concentration Versus Time Curve from 0 to the Last Measurable Concentration (AUC0-t) | Hour 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 after administration.
  Plasma concentrations of TNP-2198 were measured by a specific and validated assay. Plasma PK parameters of TNP-2198 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Maximum Observed Plasma Concentration (Cmax) of TNP-2198 | Hour 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 after administration.
  Plasma concentrations of TNP-2198 were measured by a specific and validated assay at specified time points

CONTACTS AND LOCATIONS:
Overall Officials: TenNor Clinical Trials, Study Director — TenNor
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Liu Y, Wang M, Gao L, Liu J, Zhang H, Wu M, Chen H, Lou J, Wang J, Chen J, Geng G, Ma Z, Ding Y. Safety, pharmacokinetics, and efficacy of rifasutenizol, a novel dual-targeted antibacterial agent in healthy participants and patients in China with Helicobacter pylori infection: four randomised clinical trials. Lancet Infect Dis. 2024 Jun;24(6):650-664. doi: 10.1016/S1473-3099(24)00003-3. Epub 2024 Feb 12. PMID 38359854